CLINICAL TRIAL: NCT02424838
Title: Randomized Trial Examining the Relationship Between Procedural Technique and Specimen Evaluation Methods in Patients Undergoing Endoscopic Ultrasound (EUS)-Guided Fine Needle Aspiration (FNA) of Pancreatic Masses
Brief Title: 22 G - 25 G SINS Trial for Pancreatic Masses
Acronym: SINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 618366
Record Dates: First submitted 2015-02-11; First posted 2015-04-23 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 22 gauge with suction (Active Comparator): EUS-FNA of pancreatic masses will be performed with a 22 gauge needle using suction.
  Interventions: Procedure: EUS-FNA of pancreatic masses; Device: 22 gauge needle
- 22 gauge without suction (Active Comparator): EUS-FNA of pancreatic masses will be performed with a 22 gauge needle without suction.
  Interventions: Procedure: EUS-FNA of pancreatic masses; Device: 22 gauge needle
- 25 gauge with suction (Active Comparator): EUS-FNA of pancreatic masses will be performed with a 25 gauge needle using suction.
  Interventions: Procedure: EUS-FNA of pancreatic masses; Device: 25 gauge needle
- 25 gauge without suction (Active Comparator): EUS-FNA of pancreatic masses will be performed with a 25 gauge needle without suction.
  Interventions: Procedure: EUS-FNA of pancreatic masses; Device: 25 gauge needle

INTERVENTIONS:
Procedure: EUS-FNA of pancreatic masses — EUS-FNA of pancreatic masses will be performed using a 22 or a 25 gauge needle with or without applying suction.
Device: 22 gauge needle
  Arms: 22 gauge with suction; 22 gauge without suction
Device: 25 gauge needle
  Arms: 25 gauge with suction; 25 gauge without suction

SUMMARY:
After patients have been screened and have signed informed consent, they will be taken to the endoscopy suite. Once the decision has been made to proceed with Fine Needle Aspiration (FNA), the subject will be randomized to 1 of 4 groups:

* 22 gauge (G) needle with suction
* 25 G needle with suction
* 22 G needle without suction
* 25 G needle without suction

Follow-up Phone Call Phase:

Unit staff will call patients 1 week after the procedure to check if patients had any adverse events from the procedure and this will be recorded onto the dataset.

DETAILED DESCRIPTION:
All adult patients referred to Florida Hospital for evaluation of a pancreatic mass lesion will be eligible for entry into the study. Patients will be approached at the time of procedural consent for the study.

1. After written informed consent is taken, Endoscopic Ultrasound (EUS) will be performed under conscious sedation.
2. At the time of EUS, patients who require FNA will be randomized to the two needles (22 G or 25 G needles) and to the two techniques (using suction or not using suction).
3. Computer-generated randomization assignments using the block randomization method will be obtained from the statistician prior to study enrollment. These will be placed in sequentially numbered sealed opaque envelopes and opened by the endoscopy nurse immediately after the decision to perform FNA is made. The randomization sequence will specify the needle size to be used and whether or not suction will be applied for FNA.
4. FNA will be performed in the standard fashion using one of the designated needle sizes (using the fanning technique to pass the needle 12-16 times into the lesion) by one of the experienced endosonographers in the unit. The needle stylet will be left in place for the first pass and then removed for subsequent passes. Suction will be applied during aspiration of the mass as dictated by the randomization sequence.
5. First two passes will be performed to obtain tissue sample for cell block analysis. Therefore, the tissue obtained with the first and second passes will be expressed onto a slide and into test tubes for cell block analysis.
6. From the third pass onwards, the aspirate obtained will be examined onsite by the cytopathologist, who will be available to interpret the slides immediately to determine diagnostic adequacy of the sample per standard practice. Once the diagnosis is made and the adequacy of the sample is affirmed by the cytopathologist, the procedure will be stopped and the echoendoscope will be withdrawn from the patient.
7. Total number of passes to obtain a diagnostic cytological aspirate made will be recorded at the time of procedure, as well as the occurrence of needle dysfunction, technical failure, and any immediate complications.
8. The samples taken will be transported to the pathology lab (per standard practice) where the cellular aspirate and cell block samples will be evaluated by the pathologist. 10% of samples from each subgroup (i.e. 22G with suction, 22G without suction, 25G with suction, 25G without suction) will be further analyzed for the presence of molecular markers for malignancy.
9. After the appropriate observations are deemed satisfactory, patients will be discharged as per unit policy.
10. Unit staff will call patients 1 week after the procedure to check if patients had any adverse events from the procedure and this will be recorded onto the dataset.

ELIGIBILITY:
Inclusion Criteria:

1. All patients referred to Florida Hospital Endoscopy Unit for assessment of pancreatic mass lesions that require FNA
2. Age ≥ 19 years

Exclusion Criteria:

1. Age <19 years
2. Unable to safely undergo EUS for any reason
3. Coagulopathy (INR >1.6, Thrombocytopenia with platelet count <80,000/ml)
4. Unable to provide consent for any reason
5. Pregnancy (confirmed with Standard of Care urine pregnancy test for all women with child-bearing potential)

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2014-07-28 (Actual); Primary Completion 2016-04-03 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of diagnostic cell block specimens obtained according to needle size and the use of suction. | 7 days (cell block processing in lab)
  The use of suction and a larger gauge needle during EUS-FNA is likely to increase the diagnostic yield of cell block. This may in turn translate to improved diagnosis and hence expedite patient management

SECONDARY OUTCOMES:
Diagnostic adequacy of FNA cytology | 24 hours
  1. Diagnostic adequacy of FNA cytology samples and comparison between the two needle sizes and the effect of application of suction
Median number of passes to diagnosis | 24 hours
  2. Median no. of passes required to obtain diagnostically adequate cytological samples, and comparison between the two needle sizes and suction vs. no suction
Specimen bloodiness | 24 hours
  3. Specimen bloodiness and comparison between the two needle sizes and two techniques (with and without suction)
Rate of needle dysfunction | 24 hours
  4. Rate of needle dysfunction and technical failure, and comparison between the two needle sizes and two techniques (with and without suction)
Rate of complications | 3 days
  5. Rate of complications following EUS-FNA, and comparison between the two needle sizes and two techniques (with and without suction)

CONTACTS AND LOCATIONS:
Overall Officials: Shyam S Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Participant Data.

REFERENCES:
- [Derived] Bang JY, Navaneethan U, Hasan MK, Hawes R, Varadarajulu S. Endoscopic Ultrasound-guided Specimen Collection and Evaluation Techniques Affect Diagnostic Accuracy. Clin Gastroenterol Hepatol. 2018 Nov;16(11):1820-1828.e4. doi: 10.1016/j.cgh.2018.03.004. Epub 2018 Mar 11. PMID 29535060